CLINICAL TRIAL: NCT00435760
Title: Single Dose, Double-blind, Double-dummy, 3 Period Cross-over, Placebo Controlled Clinical Trial to Assess the Reate of Onset of Action of Inhaled Aclidinium Bromide 200µg Compared to Placebo and Tiotropium 18µg in Patients With Chronic Obstructive Pulmonary Disease (COPD).
Brief Title: Clinical Trial to Assess Rate of Onset of Bronchodilator Action in Severe Stable Chronic Obstructive Pulmonary Disease (COPD) Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: M/34273/24; 2005-005804-17 (EudraCT Number)
Record Dates: First submitted 2007-02-14; First posted 2007-02-15 (Estimated); Last update posted 2016-11-17 (Estimated); Status verified 2016-11

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
Keywords: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — aclidinium bromide; Tiotropium Bromide

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- Tiotropium (Active Comparator): 1 puff, 1 day treatment
  Interventions: Drug: Tiotropium
- Placebo (Placebo Comparator): Tiotropium or Aclidinium Placebo, 1 day treatment
  Interventions: Drug: Placebo Tiotropium; Drug: Placebo LAS34273
- Aclidinium bromide (Experimental): 200 micrograms, once daily, 1 day treatment
  Interventions: Drug: Aclidinium bromide

INTERVENTIONS:
Drug: Aclidinium bromide — 200 micrograms, once daily, 1 day treatment
  Arms: Aclidinium bromide
Drug: Placebo Tiotropium — 1 puff once daily, 1 day treatment
  Arms: Placebo
Drug: Tiotropium — 1 puff of 18 µg (22.5 µg tiotropium bromide monohydrate) in the morning between 8:00 and 10:00
  Arms: Tiotropium
Drug: Placebo LAS34273 — 1 puff, 1 dat treatment
  Arms: Placebo

SUMMARY:
This trial evaluates the rate of onset of bronchodilator action of aclidinium bromide compared to placebo and tiotropium in patients with severe COPD after a single dose treatment.

DETAILED DESCRIPTION:
This is a single dose, randomised, double-blind, double-dummy, 3 period cross-over, placebo controlled, multinational, multicentre trial.

ELIGIBILITY:
Inclusion Criteria:

* Males and females aged ≥ 40 years
* Current or ex-smokers of ≥ 10 pack-year
* Clinical diagnosis of severe stable COPD

Exclusion Criteria:

* History or current diagnosis of asthma, allergic rhinitis, or atopy
* Respiratory tract infection or acute COPD exacerbation in the last 6 weeks
* Hospitalised for an acute COPD exacerbation in the last 3 months
* Evidence of contraindicated use of anticholinergic drugs

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Actual)
Dates: Start 2007-02; Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
FEV1 Percentage Increase | 30 minutes
  Percentage of patients achieving a FEV1 increase from baseline equal to or greater than 10% at 30 minutes

SECONDARY OUTCOMES:
Normalised Area FEV1 AUC 0-3h | 0-3 hours
  Normalised area under the curve (AUC) 0-3 hours of FEV1 and change form baseline in FEV1 at 30 min

CONTACTS AND LOCATIONS:
Overall Officials: Esther Garcia, MD, Study Director — AstraZeneca
Locations (1):
- Respiratory Clinical Trials Ltd, London, United Kingdom

REFERENCES:
- See also: Sponsor web site — http://www.almirall.com/webcorp2/cda/ImD_04_02.jsp
- See also: Co-Sponsor web site — http://www.frx.com
- See also: CSR Synopsis — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=4055&filename=Synopsis-m-34273-24-Final.pdf